CLINICAL TRIAL: NCT06340906
Title: Electroacupuncture in Symptom Management After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Oliver Eng, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4573; UCI 23-29 (Other: CFCCC)
Record Dates: First submitted 2024-02-27; First posted 2024-04-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective pilot/feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Each participant will attend a total of 8 treatment visits (one visit per week), over the course of 8 weeks. Each EA session will be approximately 1 hour. Participants in the treatment arm will receive EA at 10 standardized acu-points that were chosen for their therapeutic effects.
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — EA at 10 standardized acu-points that were chosen for their therapeutic effects: Zhongwan (CV12), Guanyuan (CV4), Neiguan (PC6), Shenmen (HT7), Hegu (LI4) bilateral, Zusanli (ST36), Sanyinjiao (SP6), Zhaohai (KI6), Taichong (LR3) bilateral, Tian Shu (ST25) bilateral.

SUMMARY:
The investigators are conducting this research study is to evaluate the feasibility (recruitment, compliance, safety, and acceptance) of using electroacupuncture (EA) to manage complex symptoms such as pain, nausea/vomiting, diarrhea, and insomnia in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy. Additionally, the investigators are aiming to determine the effectiveness of EA in reducing these symptoms, and to examine how EA impacts important biomarkers, or proteins in the blood, that can be used as indicators or signs of these symptoms.

DETAILED DESCRIPTION:
This is a single-arm, prospective pilot/feasibility study. Patients can be enrolled at any time prior to undergoing surgery. The protocol and interventions are as described in the above schema. Baseline assessments including the above surveys and inflammatory markers will be obtained at the preoperative visit. The same assessments will be performed at approximately 1 month s/p Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy. Electroacupuncture interventions will be performed between postoperative months 1 to 3; a total of 8 weekly interventions will be performed. A completion assessment will be performed at approximately 6 months s/p Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy.

Our specific aims are as follows:

To examine the feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy.

To characterize symptoms experienced by patients during recovery from Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy.

To evaluate the utilization of EA in symptom management during recovery from Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy.

To evaluate levels of biomarkers such as circulating brain-derived neurotrophic factor, pro-inflammatory cytokines (IL-1beta, IL-4, IL-6, IL-8, IL-10, Tumor necrosis factor-alpha), mitochondrial DNA after Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy and with utilization of EA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known peritoneal disease who are scheduled to undergo Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
* Age ≥18 years
* Eastern Cooperative Oncology Group performance status ≤2
* Patients must have adequate organ and marrow function as defined through laboratory tests
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better (class 2B is defined as having cardiac enlargement but no history of congestive heart failure)
* Expected survival greater than 9 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with coexistence of another untreated malignant neoplasm other than basal cell carcinoma of the skin within the last five years
* Sites of metastases other than loco-regional lymph nodes and peritoneum (ex. Visceral metastases such as liver, lungs, bone, brain)
* Patients with uncontrolled intercurrent illness
* Severe needle phobia
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Known bleeding disorder (e.g. hemophilia, Von Willebrand's disease, thrombocytopenia)
* Pacemaker or other electronic metal implants
* Epilepsy
* Received acupuncture therapy within the past 3 months prior to study enrollment
* Patients who are breastfeeding, pregnant or are planning get pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Number of Patients Recruited | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through the number of participants recruited (% of target recruitment).
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Patient Recruitment Rate | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through assessing the number of patients recruited per month.
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Reasons for Abstaining from Participation | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through assessing the reasons both active and potential participants declined participation.
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Recruitment Duration | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through the time spent on recruitment, in minutes.
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Number of Completed Electroacupuncture Sessions | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through patient adherence to the study procedures through assessing the number of electroacupuncture sessions successfully completed in total.
Feasibility in utilizing an EA for patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - Proportion of Completed Electroacupuncture Sessions | Through study completion; approximately 1.5 years.
  The feasibility of utilizing an EA protocol in patients who have undergone Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy will be assessed through patient adherence to the study procedures through assessing the proportion of participants completing all the scheduled electroacupuncture sessions.

SECONDARY OUTCOMES:
Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Symptoms - EORTC QLQ-C30 | All the mean scores will be compared at baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-30) is a validated questionnaire developed to assess cancer patients' health-related quality of life. It incorporates 5 functional scales (cognitive, emotional, physical, role, and social), symptom scales (e.g. pain, fatigue, insomnia), and a global health scale. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale. Higher scores represent a better global health status and better degree of functioning while lower symptom scores indicate less severe symptoms.
  In addition to this questionnaire, patients' clinical notes will be reviewed to better characterize the respective symptoms.
Efficacy of EA in managing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Symptoms - EORTC QLQ-C30 | All the mean scores will be compared at baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-30) is a validated questionnaire developed to assess cancer patients' health-related quality of life. It incorporates 5 functional scales (cognitive, emotional, physical, role, and social), symptom scales (e.g. pain, fatigue, insomnia), and a global health scale. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale. Higher scores represent a better global health status and better degree of functioning while lower symptom scores indicate less severe symptoms.
Efficacy of EA in managing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Symptoms - FACT-Cog version 3 | All the mean scores will be compared at baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  All subjects will complete the FACT-Cog version 3 questionnaire to assess self-perceived subjective cognitive function. FACT-Cog is a validated questionnaire containing 33 items in the domains of concentration, functional interference, mental acuity, memory, multitasking and verbal fluency. Total score is calculated by summing scores from all the items and ranges from 0-148, and higher scores represent better subjective cognitive functioning.
Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Symptoms - FACT-Cog version 3 | All the mean scores will be compared at baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  All subjects will complete the FACT-Cog version 3 questionnaire to assess self-perceived subjective cognitive function. FACT-Cog is a validated questionnaire containing 33 items in the domains of concentration, functional interference, mental acuity, memory, multitasking and verbal fluency. Total score is calculated by summing scores from all the items and ranges from 0-148, and higher scores represent better subjective cognitive functioning.
  This questionnaire will be utilized to better characterize the effects Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy on cognitive function. of In addition to this questionnaire, patients' clinical notes will be reviewed for more robust characterization of the symptoms.

OTHER OUTCOMES:
Biomarkers - Plasma (pg/mL) | Blood biomarkers will be measured at baseline, 1 month post-surgery, and 6 months post-surgery.
  To evaluate levels of biomarkers such as circulating brain-derived neurotrophic factor, pro-inflammatory cytokines (IL-1beta, IL-4, IL-6, IL-8, IL-10, Tumor necrosis factor-alpha), mitochondrial DNA after Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy and with utilization of EA.
Vital Signs - Blood Pressure (mmHg) | Blood pressure will only be measured at baseline.
  The systolic and diastolic blood pressure of each patient will be measured prior to surgery as part of the screening process for eligibility for participation. This is to ensure the patient's stability in both undergoing the surgery and EA.
Vital Signs - Heart Rate (bpm) | Heart rate will only be measured at baseline.
  The heart rate of each patient will be measured prior to surgery as part of the screening process for eligibility for participation. This is to ensure the patient's stability in both undergoing the surgery and EA.
Vital Signs - Body Temperature (C) | Body temperature will only be measured at baseline.
  The body temperature of each patient will be measured prior to surgery as part of the screening process for eligibility for participation. This is to ensure the patient's stability in both undergoing the surgery and EA.
Vital Signs - Respiration Rate (breaths/minute) | Respiration rate will only be measured at baseline.
  The respiration rate of each patient will be measured prior to surgery as part of the screening process for eligibility for participation. This is to ensure the patient's stability in both undergoing the surgery and EA.
Vital Signs - Oxygen Saturation Rate (%) | Oxygen saturation rate will only be measured at baseline.
  The oxygen saturation rate of each patient will be measured prior to surgery as part of the screening process for eligibility for participation. This is to ensure the patient's stability in both undergoing the surgery and EA.
Height (feet and inches) | Height will only be measured at baseline.
  The participant's height will be measured prior to surgery to ensure anesthesia dosage required for the procedure is accurate to prevent any associated risk of complications during the surgery.
Weight (kg) | Weight will only be measured at baseline.
  The participant's weight will be measured prior to surgery to ensure anesthesia dosage required for the procedure is accurate to prevent any associated risk of complications during the surgery.
Incidence of Treatment-Emergent Adverse Events - Safety Monitoring | Through study completion; Approximately 1.5 years
  Participants will be monitored for adverse events such as bruising, pain or discomfort, bleeding and possible infections. Severity are graded according to the Common Terminology Criteria for Adverse Events V5.
Biomarkers - Plasma BDNF (pg/ml) | Baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  Plasma brain-derived neurotropic factor (BDNF) levels at each time point, and changes from baseline.
Biomarkers - Plasma cytokines (IL-1β, IL-4, IL-6, IL-8, IL-10, TNF-alpha, pg/mL) | Baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  Plasma cytokine levels at each time point, and changes from baseline.
Mitochondrial DNA content | Baseline (before surgery), 1 month post-surgery, and 6 months post-surgery.
  Mitochondrial DNA (mtDNA) content at each time point, and changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Eng, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - UCI Health Susan Samueli Integrative Health Institute, Irvine, California
  - University of California Irvine, Health, Orange, California

REFERENCES:
- [Background] Lutgendorf SK, Andersen BL. Biobehavioral approaches to cancer progression and survival: Mechanisms and interventions. Am Psychol. 2015 Feb-Mar;70(2):186-97. doi: 10.1037/a0035730. PMID 25730724
- [Background] Osann K, Wilford J, Wenzel L, Hsieh S, Tucker JA, Wahi A, Monk BJ, Nelson EL. Relationship between social support, quality of life, and Th2 cytokines in a biobehavioral cancer survivorship trial. Support Care Cancer. 2019 Sep;27(9):3301-3310. doi: 10.1007/s00520-018-4617-z. Epub 2019 Jan 5. PMID 30612237
- [Background] Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA. Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol. 2003 Oct 15;21(20):3737-43. doi: 10.1200/JCO.2003.04.187. PMID 14551293
- [Background] Quenet F, Elias D, Roca L, et al: A UNICANCER phase III trial of hyperthermic intra-peritoneal chemotherapy (HIPEC) for colorectal peritoneal carcinomatosis (PC): PRODIGE 7. [Internet]. J Clin Oncol 36:LBA3503-LBA3503, 2018Available from: https://doi.org/10.1200/JCO.2018.36.18_suppl.LBA3503
- [Background] Kaya H, Sezgi C, Tanrikulu AC, Taylan M, Abakay O, Sen HS, Abakay A, Kucukoner M, Kapan M. Prognostic factors influencing survival in 35 patients with malignant peritoneal mesothelioma. Neoplasma. 2014;61(4):433-8. doi: 10.4149/neo_2014_053. PMID 24645844
- [Background] Yan TD, Deraco M, Baratti D, Kusamura S, Elias D, Glehen O, Gilly FN, Levine EA, Shen P, Mohamed F, Moran BJ, Morris DL, Chua TC, Piso P, Sugarbaker PH. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for malignant peritoneal mesothelioma: multi-institutional experience. J Clin Oncol. 2009 Dec 20;27(36):6237-42. doi: 10.1200/JCO.2009.23.9640. Epub 2009 Nov 16. PMID 19917862
- [Background] Stearns AT, Malcomson L, Punnett G, Abudeeb H, Aziz O, Selvasekar CR, Fulford PE, Wilson MS, Renehan AG, O'Dwyer ST. Long-term Quality of Life After Cytoreductive Surgery and Heated Intraperitoneal Chemotherapy for Pseudomyxoma Peritonei: A Prospective Longitudinal Study. Ann Surg Oncol. 2018 Apr;25(4):965-973. doi: 10.1245/s10434-017-6326-0. Epub 2018 Jan 8. PMID 29313146
- [Background] Bartlett EK, Meise C, Roses RE, Fraker DL, Kelz RR, Karakousis GC. Morbidity and mortality of cytoreduction with intraperitoneal chemotherapy: outcomes from the ACS NSQIP database. Ann Surg Oncol. 2014 May;21(5):1494-500. doi: 10.1245/s10434-013-3223-z. Epub 2013 Aug 29. PMID 23990289
- [Background] Low CA, Bovbjerg DH, Ahrendt S, Alhelo S, Choudry H, Holtzman M, Jones HL, Pingpank JF Jr, Ramalingam L, Zeh HJ 3rd, Zureikat AH, Bartlett DL. Depressive Symptoms in Patients Scheduled for Hyperthermic Intraperitoneal Chemotherapy With Cytoreductive Surgery: Prospective Associations With Morbidity and Mortality. J Clin Oncol. 2016 Apr 10;34(11):1217-22. doi: 10.1200/JCO.2015.62.9683. Epub 2016 Feb 22. PMID 26903574
- [Background] Ihemelandu CU, McQuellon R, Shen P, Stewart JH, Votanopoulos K, Levine EA. Predicting postoperative morbidity following cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CS+HIPEC) with preoperative FACT-C (Functional Assessment of Cancer Therapy) and patient-rated performance status. Ann Surg Oncol. 2013 Oct;20(11):3519-26. doi: 10.1245/s10434-013-3049-8. Epub 2013 Jun 8. PMID 23748607
- [Background] Moaven O, Votanopoulos KI, Shen P, Mansfield P, Bartlett DL, Russell G, McQuellon R, Stewart JH, Levine EA. Health-Related Quality of Life After Cytoreductive Surgery/HIPEC for Mucinous Appendiceal Cancer: Results of a Multicenter Randomized Trial Comparing Oxaliplatin and Mitomycin. Ann Surg Oncol. 2020 Mar;27(3):772-780. doi: 10.1245/s10434-019-08064-6. Epub 2019 Nov 12. PMID 31720933
- [Background] Morgan RB, Tun S, Eng OS: Quality of life after cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: a narrative review [Internet]. Dig Med Res 3:53-53, 2020[cited 2023 Jan 4] Available from: https://dmr.amegroups.com/article/view/6846/html
- [Background] Kuchler T, Bestmann B, Rappat S, Henne-Bruns D, Wood-Dauphinee S. Impact of psychotherapeutic support for patients with gastrointestinal cancer undergoing surgery: 10-year survival results of a randomized trial. J Clin Oncol. 2007 Jul 1;25(19):2702-8. doi: 10.1200/JCO.2006.08.2883. PMID 17602075
- [Background] Witt CM, Balneaves LG, Cardoso MJ, Cohen L, Greenlee H, Johnstone P, Kucuk O, Mailman J, Mao JJ. A Comprehensive Definition for Integrative Oncology. J Natl Cancer Inst Monogr. 2017 Nov 1;2017(52). doi: 10.1093/jncimonographs/lgx012. PMID 29140493
- [Background] Napadow V, Makris N, Liu J, Kettner NW, Kwong KK, Hui KK. Effects of electroacupuncture versus manual acupuncture on the human brain as measured by fMRI. Hum Brain Mapp. 2005 Mar;24(3):193-205. doi: 10.1002/hbm.20081. PMID 15499576
- [Background] Bao T, Patil S, Chen C, Zhi IW, Li QS, Piulson L, Mao JJ. Effect of Acupuncture vs Sham Procedure on Chemotherapy-Induced Peripheral Neuropathy Symptoms: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200681. doi: 10.1001/jamanetworkopen.2020.0681. PMID 32159808
- [Background] Chan K, Lui L, Lam Y, Yu K, Lau K, Lai M, Lau W, Tai L, Mak C, Bian Z, Zhong LL. Efficacy and safety of electroacupuncture for oxaliplatin-induced peripheral neuropathy in colorectal cancer patients: a single-blinded, randomized, sham-controlled trial. Acupunct Med. 2023 Oct;41(5):268-283. doi: 10.1177/09645284221125421. Epub 2022 Nov 3. PMID 36325677
- [Background] Wang Y, Yang JW, Yan SY, Lu Y, Han JG, Pei W, Zhao JJ, Li ZK, Zhou H, Yang NN, Wang LQ, Yang YC, Liu CZ. Electroacupuncture vs Sham Electroacupuncture in the Treatment of Postoperative Ileus After Laparoscopic Surgery for Colorectal Cancer: A Multicenter, Randomized Clinical Trial. JAMA Surg. 2023 Jan 1;158(1):20-27. doi: 10.1001/jamasurg.2022.5674. PMID 36322060